CLINICAL TRIAL: NCT03587753
Title: Understanding Liver Fat Metabolism: Studies to Understand the Role of Dietary Nutrients on Liver Fat Metabolism
Brief Title: Experiment 2: Understanding Liver Fat Metabolism
Acronym: FATOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Oxlip-2013 sub amend
Record Dates: First submitted 2018-06-20; First posted 2018-07-16 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Fatty Acid Oxidation

STUDY DESIGN:
Intervention Model Description: Randomised cross-over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unsaturated (Active Comparator): A test meal containing a unsaturated fatty acid labelled with 13C to measure hepatic fatty acid partitioning.
  Interventions: Other: Dietary fatty acid partitioning
- Saturated (Active Comparator): A test meal containing a saturated fatty acid labelled with 13C to measure hepatic fatty acid partitioning
  Interventions: Other: Dietary fatty acid partitioning

INTERVENTIONS:
Other: Dietary fatty acid partitioning — There is no intervention as such, just a physiological assessment of the partitioning and oxidation of two different types of dietary fatty acids

SUMMARY:
There is a largely unsubstantiated thought in the literature that dietary unsaturated enter oxidation pathways preferentially compared to saturated fatty acids. This study is undertaking a direct comparison of the oxidation of dietary saturated and unsaturated fatty acids.

DETAILED DESCRIPTION:
Provided subjects meet the inclusion criteria, then at least one week after the screening visit volunteers will then undertake the first two 'study days'. There will be two study days on separate occasions that will be up to 3 weeks apart. Each study day will be approximately 7 hours in duration. On each study day participants will be given a standardised 'test' meal that contains specially labelled fat molecules (stable-isotope tracer) and then repeated breath and blood samples will be taken over the course of the next 6 hours. The test meal consumed on each 'study day' will be identical in composition with only the specially labelled fat molecules being different (either unsaturated or saturated fat) and these will be given in a random order.

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent for participation in the study.

Male or Female, aged >18 and <65 years BMI >19 <35kg/m2 No medical condition or relevant drug therapy known to affect liver metabolism

Exclusion Criteria:

* • Age <18 or >65 years

  * Body mass index <19 or >35kg/m2
  * A blood haemoglobin <120mg/dL
  * Any metabolic condition or relevant drug therapy
  * Smoking
  * History of alcoholism or a greater than recommended alcohol intake
  * Pregnant or nursing mothers
  * Women prescribed hormone replacement therapy (HRT) or who have used this within the last 12 months
  * History of severe claustrophobia
  * Presence of metallic implants, pacemaker
  * Haemorrhagic disorders
  * Anticoagulant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Dietary fatty acid partitioning | 6 hours
  The appearance of the 13Clabelled fatty acid in plasma triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parry SA, Rosqvist F, Cornfield T, Barrett A, Hodson L. Oxidation of dietary linoleate occurs to a greater extent than dietary palmitate in vivo in humans. Clin Nutr. 2021 Mar;40(3):1108-1114. doi: 10.1016/j.clnu.2020.07.013. Epub 2020 Jul 22. PMID 32753348